CLINICAL TRIAL: NCT05063565
Title: An Open-Label, Prospective, Multi-Center Clinical Trial to Evaluate the Efficacy and Safety of TheraSphere™ Followed by Durvalumab (Imfinzi®) With Tremelimumab (Imjudo®) for Hepatocellular Carcinoma (HCC)
Brief Title: TheraSphere With Durvalumab and Tremelimumab for HCC
Acronym: ROWAN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2472
Record Dates: First submitted 2021-09-01; First posted 2021-10-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Carcinoma; Carcinoma, Hepatocellular; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Adenocarcinoma; Liver Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Liver Diseases
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Adenocarcinoma; Liver Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Digestive System Diseases; Liver Diseases | interventions — durvalumab; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- TheraSphere followed by Durvalumab and Tremelimumab (Experimental): TheraSphere followed by Tremelimumab plus Durvalumab administered once, then repeated administration of Durvalumab monthly up 18 months.
  Interventions: Device: TheraSphere Y-90 glass microsphere therapy; Drug: Durvalumab (Imfinzi) immunotherapy; Drug: Tremelimumab immunotherapy

INTERVENTIONS:
Device: TheraSphere Y-90 glass microsphere therapy — TheraSphere Y-90 glass microsphere therapy administered through the hepatic artery at index procedure.
Drug: Durvalumab (Imfinzi) immunotherapy — 1500 mg, every 4 weeks that continues for a maximum duration of 18 months or until confirmed progression (by site assessment), unacceptable toxicity, study withdrawal, or study early termination by the sponsor. Treatment beyond confirmed radiographic progression is permitted per patient consent if the following criteria are met:
  * Absence of clinical symptoms or signs indicating clinically significant disease progression
  * No decline in performance status
  * Absence of rapid disease progression or threat to vital organs or critical anatomical sites (i.e. new CNS metastasis, respiratory failure due to tumor compression, spinal cord compression) requiring urgent alternative medical intervention
  * No other treatment discontinuation criteria are met
Drug: Tremelimumab immunotherapy — 300 mg, single administration

SUMMARY:
The objective of the ROWAN clinical study is to assess the efficacy of local tumor control in HCC patients who receive TheraSphere followed by durvalumab and tremelimumab.

DETAILED DESCRIPTION:
A global open-label, prospective, multi-center Phase II trial designed to assess the safety and efficacy of TheraSphere administered before initiation of Durvalumab with Tremelimumab in HCC patients who are not a candidate for resection, thermal ablation or liver transplant at the time of study entry.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be aged ≥18 years at the time of screening.
2. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and accountability Act in the US, European Union (EU) data privacy regulations in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
3. Life expectancy ≥6 months.
4. HCC, diagnosed by radiographic imaging or histology.
5. Patient not a candidate for liver resection, thermal ablation, or transplantation at the time of study entry.
6. ECOG 0 or 1
7. Measurable disease by mRECIST criteria (e.g. ≥10mm of enhancement).
8. Tumor volume ≤35% of whole liver volume (determined by imaging).
9. Future liver remnant volume (FLRV) ≥30% of whole liver volume. FRLV is the volume of liver not planned to be treated with TheraSphere and free of HCC.
10. Dosimetry criteria for tumor(s) and normal tissue can be determined.
11. Patients with previous liver resection or ablation ≥6 months from end of previous treatment to TheraSphere administration.
12. Previous transarterial chemoembolization (TACE) is permitted if:

    1. Previous TACE performed ≥8 months before TheraSphere administration and
    2. Result of previous TACE was CR and
    3. Current tumor is not a recurrence of previously treated lesion
13. Patients with portal vein thrombosis (PVT) Vp0, Vp1, or Vp2.
14. Patients with HBV or HCV infection are to have documented virology status of hepatitis as confirmed by HBV and HCV serology test:

    1. Patients with HBV infection: HBV DNA load should be ≤2000 IU/mL obtained within 42 days prior to initiation of study treatment, and Anti-HBV treatment (per local standard of care; e.g., entecavir) for a minimum of 14 days prior to study entry and willingness to continue treatment for the length of the study
    2. Patients with chronic HCV infection are allowed in the study: for untreated patients, AST/ALT should be ≤3xULN and for treated patients, antiviral treatment (per local standard of care) should be stopped for a minimum of 14 days prior to study entry and AST/ALT should be ≤3xULN
15. Patients with Human Immunodeficiency Virus (HIV) infection are eligible, provided the HIV infection is well controlled with no current or previous AIDS-related complications and CD4+ T-cell (CD4+) counts ≥ 350 cells/uL
16. Negative serum pregnancy test in females of childbearing potential.
17. Adequate contraception for the patient and his/her sexual partner.
18. Adequate renal and marrow function as defined below:

    1. Hemoglobin (hgB) ≥9.0 g/dL
    2. Absolute neutrophil count (ANC) ≥1.5 x 109/L
    3. Platelet count ≥75 x 109/L
    4. Measured or calculated creatinine clearance ≥45 mL/min as determined by Cockcroft-Gault (using actual body weight)
19. Absolute lymphocyte count ≥0.5 X 109/L
20. Adequate liver function, as defined by

    1. Child-Pugh A
    2. Albumin-bilirubin (ALBI) score 1 or 2 with upper limit for ALBI score ≤ -2. Patients with confirmed Gilbert's syndrome may not have an evaluable bilirubin value; therefore, ALBI score should not be considered for such patients. Patients with Gilbert's syndrome will be eligible with any bilirubin value, as long as Albumin level is ≥ 34 g/L.
    3. AST and ALT <3 x ULN.
21. Body weight >30 kg and BMI ≥18 kg/m2.

Exclusion Criteria:

1. Any contraindication to angiography or selective visceral catheterization.
2. Cone Beam CT (CBCT) or Technetium-99m macroaggregated Albumin (99mTc-MAA) hepatic arterial perfusion scintigraphy shows any deposition to the gastrointestinal tract that may not be corrected by angiographic techniques.
3. 99mTc-MAA hepatic arterial perfusion scintigraphy shows poor tumor and/or portal vein thrombosis (PVT) targeting that would lead to a dose that does not meet the liver dosing criteria.
4. Shunting of blood to the lungs that could result in delivery of >30 Gy to the lungs in a single treatment or >50 Gy cumulative dose to the lungs in case of multiple TheraSphere treatments, as seen on 99mTc-MAA hepatic arterial perfusion scintigraphy.
5. Vp3, Vp4, hepatic vein invasion, or inferior vena cava (IVC) invasion
6. Extrahepatic metastases (patients with extrahepatic spread [EHS]):

   1. EHS is any extrahepatic lesion that, according to clinical symptoms, histology, or imaging data, is highly suspicious of being metastases.
   2. For patients with bone pain/neurological symptoms (deficit, seizure or else) at baseline and suspected of metastases at screening, a bone scan/brain MRI is recommended prior to study entry.
   3. Extrahepatic non-target non-measurable lesions (<1 cm per RECIST 1.1) are acceptable if considered not suspicious by the investigator.
7. Any previous systemic HCC treatment
8. Prior exposure to immune mediated therapy for other disease, such as other anti-PD- 1, anti-PDL-1, anti-PDL-2, anti-CTLA-4, antibodies, etc.
9. Previous liver radiation (external beam radiation therapy (EBRT) or peptide receptor radionuclide therapy (PRRT)).
10. Concurrent treatment for HCC or treatment in the last 4 weeks in another clinical study, unless it is an observational study (non-interventional) or during a non-interventional follow-up stage of an interventional study, or prior inclusion in this study
11. Hepatic encephalopathy present at study entry and/or episodes of encephalopathy (Grade ≥ 2) within 6 months prior to study inclusion.
12. HCC with infiltrative disease that is not evaluable by mRECIST.
13. Pulmonary insufficiency (defined by an arterial oxygen pressure (PaO2) of <60 mmHg, or oxygen saturation (SaO2) of <90% (Roussos & Koutsoukou, 2003) or clinically evident chronic obstructive pulmonary disease (COPD)).
14. Medical history of radiation pneumonitis or recent pneumonitis, regardless of causality
15. History of any organ allograft, including bone marrow allo and autograft.
16. History of active primary/acquired immunodeficiency, that makes patients unsuitable for additional immunotherapy in this study (per investigator and as detailed in exclusion criterion #18).
17. Active or prior documented autoimmune or inflammatory disorders (including but not limited to, inflammatory bowel disease [e.g. ulcerative colitis or Crohn's disease], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g. following Hashimoto's syndrome) stable on hormone replacement therapy
    3. Any chronic skin condition that does not require systemic therapy.
    4. Patients without active disease in the last 5 years may be included but only after consultation with the Sponsor Study physician.
    5. Patients with celiac disease controlled by diet alone.
18. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g. intra-articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
    3. Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication).
19. History of gastrointestinal bleeding within 42 days prior to study inclusion, active GI bleeding and any bleeding diathesis or coagulopathy that is not correctable by usual therapy or hemostatic agents (e.g. closure device). Patients with known varices that have not bled or which have been clinically addressed can enter the study. No endoscopic exploration is required before study inclusion.
20. Presence of biliary stent or sphincterotomy within one year prior to study inclusion.
21. History of malignancy, other than HCC, within three years, except the condition is one of the following:

    1. Adequately treated carcinoma in situ of the cervix, early squamous cell carcinoma or basal cell carcinoma of the skin, localized prostate cancer, breast ductal carcinoma in situ, or low-grade endometrial carcinoma with no myometrial invasion
    2. Localized prostate cancer under active surveillance.
    3. Other cancer when there is a negligible risk of recurrence or progression or death (5-year OS rate > 90%).
22. Major surgical procedure (as defined by the Investigator) within 42 days prior to study inclusion.
23. A history of severe allergy or intolerance to contrast agents, narcotics, sedatives or atropine that cannot be managed medically.
24. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients that cannot be managed medically.
25. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), HBV and HVC co-infection, HBV and Hep D co-infection, human immunodeficiency virus (HIV 1/2 antibodies) plus HCV or HBV co-infection.
26. Receipt of live attenuated vaccine within 30 days prior to the first dose of durvalumab and/or tremelimumab. Note: patients, if enrolled, should not receive live vaccine whilst receiving durvalumab and/or tremelimumab and up to 30 days after the last dose of durvalumab and/or tremelimumab.
27. Female patients who are pregnant or breastfeeding and who do not want to stop breastfeeding. Male or female patients of reproductive potential who are not willing to employ any effective birth control method from screening and for at least 90 days after TheraSphere administration, 90 days after the last dose of durvalumab, and 6 months after the last dose of tremelimumab.
28. Unstable chronic disease or evidence of any disease or condition that would place the patient at undue risk and preclude safe use of TheraSphere, durvalumab and tremelimumab treatment as deemed by the site principal investigator.
29. Patients who are not able to follow the TheraSphere, durvalumab or tremelimumab treatment requirements.

    For France Patients Only
30. Persons deprived of their liberty by a judicial or administrative decision, persons subject to psychiatric care under articles L. 3212-1 and L. 3213-1 who are not covered by the provisions of Article L. 1121-8 and persons admitted to a health or social establishment for purposes other than research, including:

    1. Pregnant, parturient, breast-feeding women (see also inclusion criterion 16 and exclusion criterion 27)
    2. Minors (see also inclusion criterion 1)
    3. Persons receiving psychiatric treatment (see also exclusion criteria 28)
    4. Persons admitted to a health or social establishment for purposes other than research
    5. Person of full age under curatorship
    6. Adult subject to a mandate for future protection, a family authorization, or a guardianship measure
    7. Person not affiliated or not beneficiary of a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Start of Treatment (Day 1) up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated)
  Complete response and partial response evaluated by mRECIST.

SECONDARY OUTCOMES:
Number of immune mediated AEs and SAEs. | Treatment Day 1 up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Number of patients whose durvalumab and/or tremelimumab treatment was temporarily halted, postponed or permanently discontinued due to an AE. | Treatment Day 1 up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Change from baseline in liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], gamma-glutamyl transpeptidase [GGT], alkaline phosphatase [ALK], bilirubin, albumin). | Baseline up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Change from baseline in Child-Pugh score. | Baseline up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
  Minimum value is 5 (better) and maximum value is 15 (worse).
Change from baseline in Albumin Bilirubin (ALBI) score. | Baseline up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
  Minimum value is 1 (better) and maximum value is 3 (worse).
Change from baseline in Eastern Cooperative Oncology Group (ECOG) score. | Baseline up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
  Minimum value is 0 (better) and maximum value is 5 (worse).
ORR according to localized mRECIST and RECIST 1.1. | Start of Treatment (Day 1) up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is Treated ).
DoR according to mRECIST, localized mRECIST, and RECIST 1.1. | Time of response up to progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Disease Control Rate (DCR) according to localized mRECIST, mRECIST, RECIST 1.1. | Start of Treatment (Day 1) up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is Treated).
Duration of disease control (DoDC) according to localized mRECIST, mRECIST, RECIST 1.1. | Time of disease control up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Time to best response (CR or PR) according to localized mRECIST, mRECIST, RECIST 1.1. | Start of Treatment (Day 1) up to best response (CR or PR), subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Complete response rate (CRR) according to localized mRECIST, mRECIST, RECIST 1.1. | Start of Treatment (Day 1) up to complete response, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Duration of complete response (DoCR) according to localized mRECIST, mRECIST, RECIST 1.1. | Time of complete response up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Hepatic time to progression (hTTP) according to mRECIST, RECIST 1.1. | Start of treatment (Day 1) up to hepatic progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Time to progression (TTP) according to localized mRECIST, mRECIST, RECIST 1.1. | Start of treatment (Day 1) up to progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Progression free survival (PFS) according to localized mRECIST, mRECIST, RECIST 1.1; this will include an evaluation of the PFS rate at 6, 12, 18 and 24 months. | Start of treatment (Day 1) up to progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Hepatic progression free survival (hPFS) by mRECIST, RECIST 1.1. | Start of treatment (Day 1) up to hepatic progression, subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Overall survival (OS). | Start of treatment (Day 1) up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Disease Specific Survival (DSS) | Start of treatment (Day 1) up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Proportion of patients receiving subsequent treatment for HCC after study treatment, and type of HCC treatment received. | Start of treatment (Day 1) up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Proportion of patients to undergo curative therapy (transplantation or resection). | Start of treatment (Day 1) up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Time to subsequent HCC treatment (local or systemic therapy). | Start of treatment (Day 1) up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Reason for starting subsequent HCC treatment. | Start of treatment (Day 1) up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Alpha fetoprotein (AFP) response. | Baseline up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Change from baseline in quality of life (QoL) by FACT-Hep. | Baseline up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Change from baseline in QoL by EQ-5D. | Baseline up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Pre-treatment volumes and absorbed doses to the following volumes of interest (VOIs) using 99mTc-MAA SPECT/CT imaging and Simplicit90Y dosimetry software will be determined. | Baseline Visit
  Only tumor ≥3cm of longest diameter should be considered for dosimetry assessment.
  a. Tumoral VOIs i. All Tumor(s) ii. Target lesion(s) according to mRECIST b. Perfused Liver VOI c. Normal liver tissue VOIs i. Perfused normal tissue ii. Whole liver normal tissue
Post-treatment volumes and absorbed doses to the following volumes of interest (VOIs) using Y-90 PET imaging and Simplicit90Y dosimetry software will be determined. | Treatment Visit
  Only tumor ≥3cm of longest diameter should be considered for dosimetry assessment.
  a. Tumoral VOIs i. All Tumor(s) ii. Target lesion(s) according to mRECIST b. Perfused Liver VOI c. Normal liver tissue VOIs i. Perfused normal tissue ii. Whole liver normal tissue
Correlation between tumoral absorbed doses in Gy, determined by 99mTc-MAA SPECT/CT, assessing impact on tumor response and, survival. | Start of treatment (Day 1) up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Correlation between normal tissue absorbed doses in Gy, determined by 99mTc-MAA SPECT/CT, assessing impact on number of Grade 3 or higher AEs and SAEs. | Start of treatment (Day 1) up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Correlation between tumoral absorbed doses in Gy, determined by Y-90 PET, assessing impact on tumor response and survival. | Start of treatment (Day 1) up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Correlation between normal tissue absorbed doses in Gy, determined by Y-90 PET, assessing impact on number of Grade 3 or higher AEs and SAEs. | Start of treatment (Day 1) up to subsequent anti-cancer therapy, participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).
Correlation between tumoral absorbed doses in Gy determined by 99mTc-MAA SPECT/CT and Y-90 PET. | Baseline up to post-treatment imaging visit.
Correlation between normal tissue absorbed doses in Gy determined by 99mTc-MAA SPECT/CT and by Y-90 PET. | Baseline up to post-treatment imaging visit.
Determination of dose volume histogram (DVH) for tumoral VOIs and normal liver tissue VOIs, using 99mTc-MAA SPECT/CT and Y-90 PET. | Baseline up to post-treatment imaging visit.
Whole liver and remnant liver volumes at baseline and follow-up imaging assessments measured using Simplicit90Y software. | Start of Treatment (Day 1) up to participant's death, opposition to data collection, lost to follow-up, or study termination (18 months after the last patient is treated).

CONTACTS AND LOCATIONS:
Overall Officials: Beau Toskich, MD, Principal Investigator — Mayo Clinic; Aiwu Ruth He, MD PhD, Principal Investigator — Georgetown University
Locations (36):
- United States (13):
  - University of Arizona- Banner Health, Tucson, Arizona
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Georgetown University, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Hospital, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University (Barnes-Jewish Hospital), St Louis, Missouri
  - Columbia University Irving Medical Center, New York, New York
  - Intermountain Health, Salt Lake City, Utah
- France (10):
  - CHU Nantes, Rennes, Cedex
  - Hôpital Beaujon, Clichy, Hauts De Seine
  - CHU Grenoble, Grenoble, Isere
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Clermont-Ferrand
  - Chu Henri Mondor, Créteil
  - Chru De Lille, Lille
  - CHU Montpellier, Montpellier
  - CHU Angers - Hôpital Hôtel Dieu, Nantes
  - CRLCC Eugene Marquis, Rennes
  - Hopital Paul Brousse, Villejuif
- Italy (3):
  - National Cancer Institute of Milan, Italy, Milan
  - IRCCS - Regina Elena Cancer Institute, Roma
  - Azienda Sanitaria Universitaria Integrata Friuli Centrale (ASU FC), Udine
- Spain (8):
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Gregorio Maranon, Madrid
  - Hospital Universitario Virgen de las Nieves, Madrid
  - Hospital. Ramon Y Cajal, Madrid
  - Hospital Universitari, Valencia
  - Clinico de Valladolid, Valladolid
- Switzerland (2):
  - University Hospital of Bern, Bern
  - University Hospital Geneva (HUG), Geneva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Boston Scientific Website ROWAN Clinical Trial Overview — https://www.bostonscientific.com/en-US/medical-specialties/interventional-radiology/interventional-oncology/therasphere/clinical-data/rowan-study.html